CLINICAL TRIAL: NCT05496257
Title: Calcium Hydroxide Versus Premixed Bioceramic Putty in Direct Pulp Capping of Primary Molars: An Equivalent Parallel Randomized Controlled Trial
Brief Title: Calcium Hydroxide Versus Premixed Bioceramic Putty in Direct Pulp Capping of Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Merrette Basem Khalaf Sedhom, Resident in Pediatric and Community Dentistry Department, Faculty of Dentistry, Assuit University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 524_1/11/2021
Record Dates: First submitted 2022-08-05; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Direct Pulp Capping

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (control): Calcium hydroxide cement (Active Comparator): Pulp capping material
  Interventions: Other: direct pulp capping in primary molars
- Group 2: Premixed bioceramic putty (Active Comparator): Pulp capping material
  Interventions: Other: direct pulp capping in primary molars

INTERVENTIONS:
Other: direct pulp capping in primary molars — caries will be removed, and if the pulps are exposed, the material will be place directly over the exposed pulp.

SUMMARY:
The trial will be conducted to evaluate and compare calcium hydroxide and premixed bioceramic putty regarding the clinical and radiographic outcomes of direct pulp capping in primary molars.

DETAILED DESCRIPTION:
The current equivalent parallel randomized controlled trial will be conducted to evaluate and compare calcium hydroxide and premixed bioceramic putty regarding the clinical and radiographic outcomes of direct pulp capping in primary molars over a 24-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical:

  1. Children categorized as class I or II according to American Society of Anaesthesiologists (ASA) scale.
  2. Children rated as no. 3 or 4 in Frankl behaviour rating scale (FBRS).
  3. Presence of a small carious or traumatic pulp exposure (1 mm or less). 2. Radiographic:

  <!-- -->

  1. Presence of at least two-thirds of root length.
  2. Normal lamina dura and periodontal ligament space.

Exclusion Criteria:

* 1. Clinical:

  1. History of spontaneous unprovoked toothache.
  2. Extensive crown destruction that preclude coronal restoration.
  3. Gingival swelling, sinus tract or other soft tissue pathology.
  4. Abnormal tooth mobility.
  5. A frank pulp exposure (i.e., greater than 1.0mm), requiring pulpotomy.
  6. No evidence of visible pulp exposure.

     2. Radiographic:

  <!-- -->

  1. Furcation/periapical radiolucency.
  2. Pathological internal/external root resorption.
  3. Absence of underlying permanent successor

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-11-02 (Estimated); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
Clinical findings | 2 year follow up
  The children will be recalled for postoperative clinical & radiographic assessments at the following intervals; six, twelve, eighteen,and twenty-four months.the treatment will be considered successful if none of the following clinical or radiographic findings is present:
  Clinical criteria:
  1. Pain.
  2. Tenderness to palpation or percussion
  3. Gingival swelling or sinus tract.
  4. Purulent exudate expressed from the gingival margin.
  5. Abnormal tooth mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Minia university, Minya, Egypt